CLINICAL TRIAL: NCT02203214
Title: Induced ACL Healing With the Ligamys Technique: a Prospective, Multicenter Observational Case Series
Acronym: Ligamys
Status: Completed | Type: Observational
Sponsor: Mathys Ltd Bettlach (Industry)
Responsible Party: Sponsor
Other Study IDs: V03_29082013
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Ligamys; ACL; healing
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ligamys: All patients treated with Ligamys can be included in the study. Patients must meet all of the inclusion criteria and none of the exclusion criteria to be enrolled.
  Interventions: Device: Ligamys

INTERVENTIONS:
Device: Ligamys — All patients are treated with Ligamys within 21 days after injury. The Ligamys implant has to be used in accordance with the instructions for use.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Ligamys technique for the treatment of acute ruptures of the anterior cruciate ligament in a multicenter routine clinical setting. To conduct a long-term follow-up of the case series as a post-market product surveillance endeavor.

DETAILED DESCRIPTION:
The Ligamys method was successfully applied in an animal study including eleven white alpine sheep. Healing of the torn ACL and a stable joint without signs of intra-articular damages or osteoarthritis three months postoperative were observed (Kohl KSSTA 2013). In a first clinical study with ten patients, the Ligamys surgical technique resulted in stable clinical and radiological healing of the torn ACL in nine patients with one re-rupture after four months. Nine patients obtained normal knee scores, reported excellent patient satisfaction, and could return to their previous levels of sporting activity (Kohl Swiss Med Wkly 2011).

The purpose of this study is to evaluate the safety and effectiveness of the Ligamys technique for the treatment of acute ruptures of the anterior cruciate ligament in a multicenter routine clinical setting. To conduct a long-term follow-up of the case series as a post-market product surveillance endeavor.

ELIGIBILITY:
Inclusion Criteria:

* Primary rupture of the anterior cruciate ligament
* Signed patient informed consent
* Willingness to present for follow-up
* Age between 18 and 50 years at the time of inclusion in the study
* Injury - surgery time interval of 21 days or less

Exclusion Criteria:

* Medical non-compliance
* Unwillingness to follow the rehabilitation programme
* Traumatic cartilage lesion requiring cartilage repair procedure (Microfracturing, MACI, ACT) or degenerative cartilage lesions (Outerbridge >ll and defect >1cm2)
* Non-repairable meniscus lesions requiring a resection of >20%
* Previous tendon removal on injured leg
* Relevant permanent medication (Steroids, cytostatic drugs, ...)
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with an acute rupture of the anterior cruciate ligament
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Knee stability and function plus safety aspects | 12 months follow-up
  Knee stability: Lachman test Knee function: Lysholm score, IKDC score Safety: ACL re-ruptures or instabilities leading to an implant removal

SECONDARY OUTCOMES:
Patient satisfaction, work absence, activity, pain and secondary degenerative changes of the knee joint | 10 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Eggli, Prof Dr med, Principal Investigator — Klinik Sonnenhof, Switzerland
Locations (3):
- UZ Gent, Ghent, Belgium
- Universitätsklinikum Münster, Münster, Germany
- Sonnenhof, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Click here for more information about this treatment option — http://www.ligamys.com